CLINICAL TRIAL: NCT06305273
Title: Effectiveness of Two Different Body Positions During Facemask Ventilation in Class 3 Obesity Patients: a Randomized Crossover Trial
Brief Title: Effectiveness of Two Different Body Positions During Facemask Ventilation in Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 23-0150-A
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized cross-over trial to be conducted at Mount Sinai Hospital (Toronto, Ontario, Canada).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine (Experimental): Participant will be ventilated with facemask while in supine position.
  Interventions: Other: Head position for face mask ventilation during induction supine
- Head elevated (Experimental): Participant will be ventilated with facemask while in head elevated position.
  Interventions: Other: Head position for face mask ventilation during induction head elevated

INTERVENTIONS:
Other: Head position for face mask ventilation during induction supine — Participant to be ventilated starting 2 minutes after induction of general anesthesia via a face mask while in supine position. Participants will be crossed over to the head elevated position after the first measurement is obtained.
  Arms: Supine
Other: Head position for face mask ventilation during induction head elevated — Participant to be ventilated starting 2 minutes after induction of general anesthesia via a face mask while in head elevated position. Participants will be crossed over to the supine position after the first measurement is obtained.
  Arms: Head elevated

SUMMARY:
It is important to provide enough oxygen to the patients who are asleep during surgery. One way to do this is by using a mask placed over the face to help them breathe. When it becomes difficult getting enough oxygen into the patient's body using the mask, it's called difficult mask ventilation. There can be different reasons for this, and having a higher BMI is one of them. Body physique is assessed by Body Mass Index (BMI). This calculation gives an indication of a person's weight relative to their height.

There is some evidence in the research literature to suggest that when the patient is positioned in a way that helps their airway, like using a device to lift their head and torso 25 degrees , it might help the process of getting enough oxygen work better. The study aims to determine if patients with high BMI can breathe better using a face mask while they are in a head elevated position compared to lying flat on their back.

DETAILED DESCRIPTION:
Facemask ventilation is an important technique applied by anesthesiologists after induction of general anesthesia and before tracheal intubation. It is also used as a rescue maneuver in situations where a patient's consciousness is compromised affecting oxygenation. Obesity is well known to be one of the difficult predictors for facemask ventilation. In fact, the occurrence of difficult facemask ventilation is more frequent in obese patients than non obese. One of the maneuvers described to optimize the effectiveness of facemask ventilation in the general population is positioning the patient in a 25 degree head elevated position. A previous study has demonstrated improvement in facemask ventilation in obese patients with BMI from 30 to 40 kg/m2 in the head elevated position, compared to supine. However, it is not yet determined if this is applicable to patients with a BMI above 40 kg/m2. Adult obese patients with BMI of at least 40 kg/m2 will be randomized to be ventilated after induction of general anesthesia via a face mask while in one of the positions: supine or head elevated, while the volume of air that enters and exits the lungs is measured. Participants will then be changed to the second position, ventilated in the same manner and measures obtained again.

Do patients with class 3 obesity positioned in the head elevated position can be better ventilated with a face mask and positive pressure, compared to the supine position?

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 kg/m2
* age > 18 years
* scheduled for elective surgery under general anesthesia
* have the ability to comprehend the rationale for the study and provide consent

Exclusion Criteria:

* pregnancy,
* risk of aspiration of gastric content
* patients using glucagon-like peptide(GLP)-1 agonists
* emergency cases
* upper airway disease or airway anatomical abnormalities
* presence of major cardiovascular, respiratory, or cerebral vascular disease
* if the provider anesthesiologist indicates an awake technique to secure the airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Average tidal volume | During induction.
  The primary outcome for this trial is the average tidal volume in 10 ventilations in each position, flat or head elevated.

SECONDARY OUTCOMES:
Predictors for difficult mask ventilation like BMI | During induction
  Secondary outcome will be: the incidence and correlation of other predictors for difficult mask ventilation like BMI.
Predictors for difficult mask ventilation like presence of beard | During induction
  Secondary outcomes will be: the incidence and correlation of other predictors for difficult mask ventilation like, presence of a beard.
Predictors for difficult mask ventilation like Mallampati classification III or IV | During induction
  Secondary outcomes will be: the incidence and correlation of other predictors for difficult mask ventilation like Mallampati classification III or IV.
Predictors for difficult mask ventilation like age of 57 yo or older. | During induction
  Secondary outcomes will be: the incidence and correlation of other predictors for difficult mask ventilation like, age of 57 yo or older.
Predictors for difficult mask ventilation like severely limited mandibular protrusion | During induction
  Secondary outcomes will be: the incidence and correlation of other predictors for difficult mask ventilation like severely limited mandibular protrusion.
Predictors for difficult mask ventilation like history of snoring. | During induction
  Secondary outcomes will be: the incidence and correlation of other predictors for difficult mask ventilation like history of snoring.
Oropharyngeal airway | During induction
  Incidence of use of an oropharyngeal airway during the protocol.
Insufficient mask ventilation | During induction.
  Incidence of insufficient mask ventilation (defined as tidal volume (Vt) < 4 ml/kg IBW), or failed facemask ventilation defined as absence of End-tidal carbon dioxide(EtCO2) after 3 consecutive ventilations.

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio Zasso, MD, Principal Investigator — MOUNT SINAI HOSPITAL